CLINICAL TRIAL: NCT05741775
Title: Efficacy of Physiotherapy Intervention Among University Students With Migraine Symptoms
Brief Title: Physiotherapy Intervention for Migraine Symptoms
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Kiruthika Selvakumar, Principle Investigator (Lecturer), Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U/SERC/188/2022
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Migraine
Keywords: Migraine symptoms; Aerobic exercise; Biofeedback training; University students
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Three groups will be present. One group receives aerobic training, second group receives biofeedback training and the last group receives patient education. So during the trial, participants in one group receive aerobic intervention "in parallel" to participants in the other group, who receive biofeedback training and patient education.
Who Masked: Participant
Masking Description: A single blinding method will be used. The participant will not know whether he or she belongs to experimental group. Only the primary researcher performing the study will know if the participants are into aerobic training, biofeedback training or control group. Single blinding will be used in this study because the results produced are less likely to be biased.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic training (Experimental): Participants in the aerobic group will undergo a training that includes walking, static bicycle, and neck exercise. The participants start the session with a warm-up for 5 minutes followed by 30 minutes of aerobic exercise and end with 5 minutes of cool-down exercise. 40 minutes/ session, 3 times per week for 6 weeks.
  Interventions: Other: Aerobic training
- Biofeedback training (Experimental): Participants in this group will undergo an electromyography (EMG) biofeedback training for trapezius and frontalis using rose for relaxation 3 times per week for 6 weeks. Each session will be for 30 minutes with a 5-minute resting period between each muscle session.
  Interventions: Other: Biofeedback Training
- Waitlist Control group (No Intervention): The control group will receive the patient education sheet with the basic information about migraine in terms of symptoms, triggers, and prevention tips. This group is also called as "waitlist control group" who will receive intervention after the active treatment group.

INTERVENTIONS:
Other: Aerobic training — The warm-up exercise will include light aerobic activity and some dynamic stretching movements. Similarly, the cool down exercises will include buttock stretch, hamstring stretch, inner thigh stretch, calf stretch and thigh stretch. Each stretch to be performed for 5 repetitions with a hold time of 15 seconds for each. An elastic band secured around the head will be used to apply local pressure over the area. Kettler Computeranleitung Advanced display will be used to train static cycling. ProAction BH Treadmill G6700 instrument will be used for aerobic training.
  Other Names: Group 1
  Arms: Aerobic training
Other: Biofeedback Training — Neurotrac myoplus 4 pro instrument will be used for EMG biofeedback training.
  Other Names: Group 2
  Arms: Biofeedback training

SUMMARY:
The goal of this randomized control trial is to analyse the effectiveness of Physiotherapy intervention among university students with migraine symptoms. The main objective is:

1. To determine the effect of aerobic exercise on the resting-state brainwaves among university students in UTAR with migraine symptoms compared with biofeedback and control exercise.
2. To analyse the influence of aerobic exercise on the sleep quality and quality of life among the cohort compared with biofeedback and control exercise.

Although the Migraine Research Foundation listed three main types of non-drug treatments for migraine are lifestyle advice, therapies, and exercises. Some common aerobic exercises such as walking, jogging, a behavioral weight loss program, cycling, and a combination of cross-training, walking, jogging, and cycling are suggested to be beneficial to the migraine patients but there remains no specific protocol established till now. Hence the other main objective of this is to establish a aerobic exercise protocol for patients with migraine symptoms.

DETAILED DESCRIPTION:
Habitual aerobic exercise has a major advantage of preventing or reducing symptoms of several chronic diseases and medical conditions. Aerobic or cardiovascular exercise by definition is a form of bodily movement that is fueled by aerobic energy-generating processes, where the energy demands of the exercise performed do not exceed the rate at which the cardiovascular system can supply oxygen to working muscles. Aerobic exercises have already proven to reduce frequency, duration, severity or associated disability in migraine. The physiology is that when one exercises, the body releases endorphins, which are the body's natural painkillers and natural anti-depressants chemicals called enkephalins. According to Centre of Disease Control and Prevention (CDC), adult should exercise 150 minutes of moderate intensity aerobic exercise and 2 or more days a week of muscle strengthening each week for relief of migraine or primary headaches. Similarly, a study conducted comparing neck treatment and aerobic exercise concluded that 5 weeks of intervention for migraine patient responded with better outcomes. According to American migraine foundation the exercise program, should include the cardiorespiratory fitness, flexibility exercises and muscular strengthening. For this reason, several studies encourage a multidisciplinary and tailored treatment approach for these patients. Hence the study aim to assess the efficacy of physiotherapy intervention especially aerobic exercise among university students with migraine symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate, and postgraduate students from Universiti Tunku Abdul Rahman
* 4 of 5 on the Migraine Screen Questionnaire

Exclusion Criteria:

* Score of more than or equal to 5 on the visual aura rating scale,
* Diagnosed to have a secondary headache (headache attributed to the causative disorder example: infection, trauma, injury to head/ or neck)
* Pregnancy,
* Took medication for neurological conditions like stroke, multiple sclerosis and took medications for cardiorespiratory conditions like asthma,
* Took medications for headache and
* Unwilling to participate will be excluded

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-09-18 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
resting-state EEG | 20 minutes
  Recording of resting-state EEG will be performed using MUSE 2 a portable EEG recording device. The headset has four dry sensors (two mastoid and two forehead sensors) and fits over the ears and extends at an angle over the middle of the forehead when properly fitted with 3 reference electrodes. Once the headband is fitted, the mind monitor app will be used for data acquisition. The data obtained will be imported to MATLAB using EEGLAB function plugins (muse monitor app) CSV file. Once imported the pre-processing steps will be done to run Independent Component Analysis (ICA). Amplitude and frequency, frequency band ratio, power spectrum density and coherence will be the primary measurement analyzed for the resting-state EEG recording,

SECONDARY OUTCOMES:
Pittsburgh Sleep index | 10 minutes
  Pittsburgh Sleep index is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. 19 individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Migraine Specific Quality of life | 10 minutes
  Migraine Specific Quality of life is a 14-item instrument that measures the impact of migraine across three essential aspects of a patient's health-related quality of life over the past 4 weeks: role function-restrictive (RR), role function-preventive (RP), and emotional function (EF). Raw dimension scores are computed as a sum of item response and rescaled from a 0 to 100 scale. The higher the score better is the quality of life.
Health survey questionnaire | 5 minutes
  Characteristics like frequency, severity and duration of migraine. Level of pain scored on a four-point numerical rating scale (0-3) equivalent to no, mild, moderate, and severe pain: 0 no pain. 1 mild pain, does not interfere with usual activities 2 moderate pain, inhibits but does not wholly prevent usual activities 3 severe pain, prevents all activities. The other components are expressed as either decreased/ increased/ remains the same/ unable to recall.

CONTACTS AND LOCATIONS:
Locations (1):
- UTAR, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol may be shared

REFERENCES:
- [Background] Santiago MD, Carvalho Dde S, Gabbai AA, Pinto MM, Moutran AR, Villa TR. Amitriptyline and aerobic exercise or amitriptyline alone in the treatment of chronic migraine: a randomized comparative study. Arq Neuropsiquiatr. 2014 Nov;72(11):851-5. doi: 10.1590/0004-282x20140148. PMID 25410451
- [Background] Varkey E, Cider A, Carlsson J, Linde M. Exercise as migraine prophylaxis: a randomized study using relaxation and topiramate as controls. Cephalalgia. 2011 Oct;31(14):1428-38. doi: 10.1177/0333102411419681. Epub 2011 Sep 2. PMID 21890526
- [Background] Wallasch TM, Kropp P. Multidisciplinary integrated headache care: a prospective 12-month follow-up observational study. J Headache Pain. 2012 Oct;13(7):521-9. doi: 10.1007/s10194-012-0469-y. Epub 2012 Jul 12. PMID 22790281
- [Background] Puledda F, Shields K. Non-Pharmacological Approaches for Migraine. Neurotherapeutics. 2018 Apr;15(2):336-345. doi: 10.1007/s13311-018-0623-6. PMID 29616493
- [Background] Parsons AA. Cortical spreading depression: its role in migraine pathogenesis and possible therapeutic intervention strategies. Curr Pain Headache Rep. 2004 Oct;8(5):410-6. doi: 10.1007/s11916-996-0016-0. PMID 15361327
- [Background] Ouyang CS, Chiang CT, Yang RC, Wu RC, Lin LC. Quantitative electroencephalogram analysis of frontal cortex functional changes in patients with migraine. Kaohsiung J Med Sci. 2020 Jul;36(7):543-551. doi: 10.1002/kjm2.12213. Epub 2020 Apr 7. PMID 32259398
- [Result] Irby MB, Bond DS, Lipton RB, Nicklas B, Houle TT, Penzien DB. Aerobic Exercise for Reducing Migraine Burden: Mechanisms, Markers, and Models of Change Processes. Headache. 2016 Feb;56(2):357-69. doi: 10.1111/head.12738. Epub 2015 Dec 8. PMID 26643584
- See also: The association between migraine and physical exercise. — http://doi.org/10.1186/s10194-018-0902-y